CLINICAL TRIAL: NCT04004585
Title: Get Up For Your Health: A Behaviour Change Intervention to Reduce Sedentary Behaviour for People With COPD
Brief Title: A Sedentary Behaviour Reduction Intervention for People With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Park Healthcare Centre (Other)
Responsible Party: Principal Investigator, Roger Goldstein, Clinical Professor, West Park Healthcare Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-012-WP
Record Dates: First submitted 2019-06-30; First posted 2019-07-02 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: COPD
Keywords: Sedentary behaviour; Behaviour change; Theoretical Domains Framework
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This was a single arm study with all participants receiving the same intervention. Participants will receive a 4-week behaviour change intervention underpinned by the Theoretical Domains Framework (TDF) that aims to reduce sedentary behaviour.
  Interventions: Behavioral: Get Up For Your Health

INTERVENTIONS:
Behavioral: Get Up For Your Health — The intervention is a 4-week behaviour change intervention underpinned by the Theoretical Domains Framework (TDF) that aims to reduce sedentary behaviour. The intervention consists of one individualized face-to-face session and 3 subsequent weekly points of contact (face-to-face meetings or phone calls).
  Behaviour change techniques will be provided including education, verbal persuasion, environmental restructuring and goal-setting.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a major cause of disability. Individuals with COPD are more likely to spend prolonged periods of time in sedentary behaviour (SB) and less in light physical activity compared to their healthy peers. SB is associated with exercise intolerance, reduced motivation to exercise, lower self-efficacy and more frequent acute exacerbations among people with COPD. To date, there is very limited information regarding behavioural approaches to reduce SB in people with COPD. The aim of this study is to examine the feasibility of a new 4-week theory-informed behaviour change intervention to reduce SB in individuals with COPD.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD confirmed by spirometry Forced expired volume to forced vital capacity ration (FEV1/FVC) less than 0.7
* An ability to ambulate.
* An ability to provide informed consent.

Exclusion Criteria:

* Presence of co-existing conditions that may prevent participation in the intervention.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | 4 weeks
  Enrollment rate is calculated as a percentage (number of people enrolled/ number of people approached)
Completion rate | 4 weeks
  Percentage of those enrolled who completed the program
Participants satisfaction | 4 weeks
  Participant satisfaction will be assessed on a percentage scale of 0 to 100, with 100 being the best possible score.
Adherence to wearing the activity monitor | 4 weeks
  Percentage of those who were able to provide data for at least 8 hours per day of wearing time during waking hours and for at least 4 days/week for the entire duration of the study

SECONDARY OUTCOMES:
Change in sedentary time | Baseline - week 4 (post-intervention)
  To assess the change in sedentary time as measured using an accelerometer from baseline to post-intervention.
Change in number of sit-to-stand transitions | Baseline - week 4 (post-intervention)
  To assess the change in the number of sit-to-stand transitions as measured using an accelerometer from baseline to post-intervention.
Change in daily number of steps | Baseline - week 4 (post-intervention)
  To assess the change in the number of steps as measured using an accelerometer from baseline to post-intervention.
Change in self-efficacy | Baseline - week 4 (post-intervention)
  To assess the change in self-efficacy to sit less using a scale adapted from the Multidimensional Self-Efficacy Scale over time from baseline to post-intervention. The scale consists of 9 items that measures 3 components of self-efficacy (task, coping and scheduling) with each item is measured on a scale of 0 (no confidence at all) up to 100 (complete confidence). The total score is the average of the scores of the 9 items.
Change in outcome expectations | Baseline - week 4 (post-intervention)
  To assess the change in the outcome expectations using a 15-item scale adapted from the Multidimensional Outcome Expectations for Exercise Scale over time from baseline to post-intervention. The questionnaire is a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree), that assesses physical outcome expectations (6 items), social outcome expectations (4 items), and self-evaluative outcome expectations (5 items) with the higher the scores the more positive the outcome expectations are. The total score is the sum of the score of the 15 items.
Change in knowledge of sedentary behaviour | Baseline - week 4 (post-intervention)
  To assess the change in sedentary behaviour using an 8-item True or False questionnaire with higher scores indicating better knowledge of sedentary behaviour

CONTACTS AND LOCATIONS:
Overall Officials: Roger Goldstein, MD, Principal Investigator — West Park Healthcare Centre; Dina Brooks, PhD, Principal Investigator — McMaster University
Locations (1):
- West Park Healthcare Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wshah A, Selzler AM, Hill K, Brooks D, Goldstein R. Embedding a Behavior Change Program Designed to Reduce Sedentary Time Within a Pulmonary Rehabilitation Program Is Feasible in People With COPD. J Cardiopulm Rehabil Prev. 2022 Jan 1;42(1):45-51. doi: 10.1097/HCR.0000000000000624. PMID 34520411